CLINICAL TRIAL: NCT00859209
Title: Capnography in Infants Ventilated With High Frequency Ventilation: Prospective, Observational, Multi-Center Study
Brief Title: Capnography in Infants Ventilated With High Frequency Ventilation
Status: Completed | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 68/08
Record Dates: First submitted 2009-02-10; First posted 2009-03-10 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2009-03

CONDITIONS: Infants in NICU Ventilated With HFV
Keywords: HVF; Premature infants; ETCO2
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that dEtCO2 measured by the Microstream® technique via a double-lumen ETT in infants ventilated with HFV would be feasible and adequately represent the arterial CO2 (PaCO2).

DETAILED DESCRIPTION:
All infants with double lumen ETT on HFV are eligible.

ELIGIBILITY:
Inclusion Criteria:

* All intubated infants with double lumen ETT ventilated with HFV

Exclusion Criteria:

* Infants ventilated with single lumen ETT

Ages: 1 Minute to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants in NICU ventilated with HFV
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The investigators primary outcome measure will be to evaluate the accuracy and the correlation of Microstream® dEtCO2 with the gold standard of PaCO2. | A Year

CONTACTS AND LOCATIONS:
Overall Officials: Kugelman Amir, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Kugelman A, Riskin A, Shoris I, Ronen M, Stein IS, Bader D. Continuous integrated distal capnography in infants ventilated with high frequency ventilation. Pediatr Pulmonol. 2012 Sep;47(9):876-83. doi: 10.1002/ppul.22524. Epub 2012 Feb 10. PMID 22328495